CLINICAL TRIAL: NCT06105060
Title: Clinical and Biochemical Study of the Effects of Rosuvastatin, Vitamin E, and N-Acetyl Cysteine on Patients With Non-alcoholic Steatohepatitis: a Randomized Controlled Trial
Brief Title: Clinical Effects of New Approach on Patients With Non-alcoholic Steatohepatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Yahia Zakaria Abu Hamza, Assistant Lecturer of Clinical Pharmacy (pharmacy practice department)Faculty of Pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Comparative study of NASH
Record Dates: First submitted 2023-10-03; First posted 2023-10-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Rosuvastain; N-Acetyl Cysteine; Vitamine E; NASH; Fibroscan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Rosuvastatin Calcium; Acetylcysteine; Vitamin E

STUDY DESIGN:
Intervention Model Description: This study will be randomized controlled, parallel and prospective 6-months duration study. Accepted patients will be randomized into 4 groups. The size of the sample is calculated using open EPI software (www.openepi.com) and according to NASH prevalence in Egypt.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Rosuvastatin group): (Active Comparator): 40 patients will receive Crestor (Rosuvastatin 20mg/day orally for 6 months).
  Interventions: Drug: Rosuvastatin 20mg
- Group 2 (N-acetyl cysteine group (NAC): (Active Comparator): 40 patients will receive high dose of NATURAL TRUTH'S NAC cap 2400 mg /day for 6 months.
  Interventions: Drug: Rosuvastatin 20mg
- Group 3 Two separate drugs ("N-acetyl cysteine" and "Rosuvastatin group"): (Active Comparator): 40 patients will receive "NAC dose 2400 mg" and "Rosuvastatin 20mg /day" for 6 months.
  Interventions: Drug: Rosuvastatin 20mg
- Group 4 (Control group): (Placebo Comparator): 40 patients will receive Vitamin E 400 mg twice daily for 6 months.
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 20mg — to evaluate and compare the protective outcomes of using Rosuvastatin, Vitamin E, and N-acetyl cysteine in Egyptian patients with NASH.
  Other Names: N-acetyl cysteine; Vitamin E

SUMMARY:
This study aims to evaluate and compare the protective outcomes of using Rosuvastatin, Vitamin E, and N-acetyl cysteine in Egyptian patients with NASH.

The primary endpoint of this 6-month study would be an improved degree of fibrosis with no worsening of NASH or NASH resolution with no worsening of fibrosis and steatosis that the study considered successful if either 1ry endpoint is met.

The secondary endpoint of this study is the improvement of biochemical markers related to steatosis, inflammation, oxidative stress, insulin resistance, and liver fibrosis.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the buildup of excessive fat in the liver without of extensive alcohol consumption and the lack of any secondary cause. The prevalence of NAFLD has risen dramatically, now affecting 20-40% of the population. NAFLD is one of the most frequent chronic liver diseases currently attributed to the rising rates of obesity and type 2 diabetes. The condition can proceed from simple steatosis to nonalcoholic steatohepatitis (NASH), characterized by hepatic damage with inflammatory infiltration, and then on to liver fibrosis, cirrhosis, and hepatocellular cancer. Currently, there is no approved drug for NASH. Consequently adjustments to lifestyle remain the mainstay of treatment despite the considerable disease burden and mortality associated predominantly with advanced diseases, i.e., NASH and fibrosis. Regarding the development of NAFLD, Despite widespread consensus on the "two hits" hypothesis linking insulin resistance (IR) and oxidative stress, the mechanism of NAFLD was thought to be highly nuanced and unexplained.

The free, un-esterified form of cholesterol appears toxic to hepatocytes, leading to inflammation and fibrosis in the liver. In particular, the steatotic liver cells form crown-like structures due to the accumulation of cholesterol crystals within the hepatocytes, which triggers an inflammatory response via activated Kupffer cells surrounding the hepatocytes. In addition, cholesterol crystals stimulate the inflammasome in Kupffer cells by activating the Nucleotide-binding oligomerization domain (NOD), leucine-rich repeats (LRR), and pyrin domain-containing protein 3 (NLRP3).

Herein, drugs known as statins block the enzyme 3-hydroxy-3-methyglutaryl coenzyme A reductase. Statins are effective medications for decreasing cholesterol and lowering the risk of cardiovascular events. Because NAFLD is characterized by free cholesterol aggregation in hepatocytes, their ability to reduce cholesterol levels is thought to be helpful. Statins also reduce the production of isoprenoids, which are byproducts of the mevalonate pathway. Isoprenoids modulate the intracellular signalling of many receptors regulating liver inflammation and fibrosis by prenylating/activating small guanosine triphosphate (GTP)ases. The significant anti-inflammatory and anti-fibrotic benefits were shown in an experimental model of NAFLD and NASH after statin-related suppression of this isoprenoid dependent mechanism.

Rosuvastatin showed promising results in enhancing liver-specific outcomes of NAFLD in preliminary investigations. Six individuals without diabetes and hypertension who were dyslipidemic and had metabolic syndrome and biopsy-proven NASH had treated with rosuvastatin 10 mg/day. After 12 months, a second biopsy and liver ultrasonography revealed that all symptoms associated with NASH (steatosis, necroinflammation, and fibrosis) had disappeared in 5 of 6 individuals. Rosuvastatin was additionally associated to a 76% and 61% decrease in ALT and AST activity, respectively. Another small prospective study with 23 NAFLD patients with dyslipidemia, rosuvastatin 10mg/day yielded similar results.

Recently, oxidative stress is characterized by an imbalance between the production and elimination of free radical species, is a hallmark of metabolic syndrome. Numerous studies have established a connection between elevated oxidative stress indicators and the development of NAFLD. Although oxidative stress is a major factor in how the liver functions in NAFLD, inflammation has also been shown to have a significant role.

Interleukin (IL)-6, tumor necrosis factor alpha (TNF-), nuclear factor kappa-light-chain-enhancer of activated B cells (NF-B), and transforming growth factor beta (TGF )-1 are pro-inflammatory mediators that, when elevated for an extended period of time, accelerate NASH and liver fibrosis.

The pharmaceutical therapies with strong antioxidant characteristics, such as N-acetyl cysteine (NAC), are crucial in reducing oxidative stress and inflammation caused by metabolic dysfunction. Its efficacy in restoring glutathione (GSH) levels in hepatocytes and decreasing pro-inflammatory cytokines has been demonstrated in animal models of nonalcoholic fatty liver disease. In a comprehensive analysis of literature published in 2015, it has been hypothesized that NAC can reduce oxidative stress and inflammation in the liver, hence enhancing its functional capacity. Since then, a plethora of studies have been published looking at NAC's effectiveness in reducing metabolic syndrome symptoms.

Vitamin E is the most abundant lipid-soluble chain-breaking antioxidant in the human body. Vitamin E family compounds are anti-atherogenic, anti-inflammatory and being powerful antioxidants.The American Association for the Study of Liver Diseases (AASLD) and the National Institute for Health and Care Excellence (NICE) recommend 800 IU of vitamin E daily for persons with biopsy-proven NASH.

NAFLD is a worldwide epidemic expected to be the leading cause of chronic liver disease in the next decade. Patients with NASH have high risk to develop liver complications such as cirrhosis, cancer, hepatic failure, morbidity and mortality. While numerous drugs have undergone clinical testing, most have shown inconsistent outcomes and have poorly tolerated side effects. Currently, there is no FDA-approved medication for the treatment of NASH. Consequently, exerting great effort is to find specific treatment for patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* All patients are diagnosed to have fatty liver grading 1, 2 or 3 on abdominal ultrasound with Hepatic steatosis index > 36 to be considered as a NAFLD patient.
* NASH diagnosis using Fibroscan detecting the degree of steatosis and fibrosis.
* NASH diagnosis is by non-invasive Scoring such as (FAST Score) Cytokeratin-18 >240 U/L Mild to moderate elevation of hepatic liver enzymes: serum aminotransferases (>2 but <5 times upper normal limit)
* Stable dietary habits and physical activity pattern.

Exclusion Criteria:

* Current or history of significant alcohol consumption.
* Use of drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins).
* Prior or planned bariatric surgery.
* Uncontrolled diabetes defined as Hemoglobin A1c 9.5% or higher.
* Evidence of other forms of chronic liver disease as Hepatitis B, Hepatitis C, Wilson's disease, Alpha-1-antitrypsin(A1AT) deficiency, Hemochromatosis, drug-induced liver disease.
* The presence of contra-indications of NAC or rosuvastatin.
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial and breast feeding.
* Use of other drugs known to have possible positive effects on steatosis.
* If there are any conditions where fibroscan could be contra-indicated. The patients refuse participating or completing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — aged ≥18 years.
Enrollment: 175 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 months
  (systolic blood pressure/diastolic blood pressure in mmHg normal blood pressure is 120/80 mmHg).
Hight | 6 months
  In meters (m) .
Weight | 6 months
  in Kilograms (kg)
Waist circumference | 6 months
  in centimeters (cm).
Body mass index (BMI) | 6 months
  The BMI calculation divides an adult's weight in kilograms (kg) by their height in meters (m) ^2. (BMI in kg/m^2).
Clinical examination | 6 months
  Abdominal ultrasound: to examine right upper quadrant pain or dullness, Mild or moderate hepatomegaly, and The appearance of a hyperechoic liver (showing more echogenicity than the kidneys), vascular blurring, and deep attenuation on ultrasonography are consistent with liver steatosis. and the appearance of bright liver)
FibroScan-AST (FAST Score): | 6 months
  Base line and at the end of the study period 3months
  * Steatosis or /and fibrosis Grade of the liver is examined by Fibroscan® of the liver tissue.
  * The FAST score was calculated using [e ˆ(- 1·65 + 1·07 × In(LSM) + 2·66∗10-8 × CAP3 - 63.3 × AST-1)]/[1 + e ˆ (- 1·65 + 1·07 × In(LSM) + 2·66∗10-8 × CAP3 - 63.3 × AST-1)] as carried out by
  Scoring system were used to determine:
  A-fibrosis staging (F0-F4). For F0-F1, LSM <7.9 kPa; for F2, LSM of 7.9 to <8.8 kPa; for F3, LSM of 8.8 to <11.7 kPa; and for F4 LSM ≥11.7 kPa. B-steatosis grade (S0-S3) to determine the presence of NAFLD. S0 was defined as a CAP <248 dB/m (<10% steatosis); S1 as CAP of 248 to <268 dB/m (10% to <33% steatosis (mild)); S2 as CAP of 268 to <280 dB/m (33% to <66% steatosis (moderate)); and S3 as CAP ≥280 dB/m (≥66% steatosis (severe))
Liver Fibrosis Index FIB-4 score (FIB-4 score): | 6 months
  Platelets count ( PLT) with FIB-4 score. The formula for FIB-4 is: Age ([yr] x AST [U/L]) / ((PLT [10(9)/L]) x (ALT [U/L])(1/2)).
  The value of FIB-4 below 1.30 is considered as low risk for advanced fibrosis. The value of FIB-4 over 2.67 is considered as high risk for advanced fibrosis. The value between 1.30 and 2.67 are considered as intermediate risk of advanced fibrosis.
Fasting blood glucose level | 6 months
  This is by venous blood sample collection in order to assess:
  Fasting blood glucose level, Normal level between 70 mg/dL and 110 mg/dL .
Homeostasis Model Assessment (HOMA-IR), | 6 months
  This is by venous blood sample collection in order to assess:
  Fasting insulin with calculation of Homeostasis Model Assessment (HOMA-IR), Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Kidney function tests: | 6 months
  This is by venous blood sample collection in order to assess:
  Serum urea ( Normal Range (NR): 5 to 20 mg/dl) Serum creatinine (NR For adult men, 0.74 to 1.35 mg/dL and For adult women, 0.59 to 1.04 mg/dL.
Lipid profile: | 6 months
  This is by venous blood sample collection in order to assess:
  Lipid profile:
  Total cholesterol ( normal level lower than 200mg/dL) High density lipoprotein cholesterol (HDL), normal level is between 40 to 60mg/dL Triglycerides, normal in range when in between 10 to 150 mg/dL. Low-density lipoprotein (normal level is between 70 to 130mg/dL).
Liver function tests: | 6 months
  This is by venous blood sample collection in order to assess:
  Alanine transaminase(ALT): The normal range is 4 to 36 U/L Aspartate aminotransferase (AST): The normal range is 8 to 33 U/L Alk. Phospatse:The normal range is 44 to 147 IU/L Gamma-glutamyl transferase (GGT): reference range for adults is 5 to 40 U/L.
Serum Malondialdehyde (MDA) level (nM): | 6 months
  This is by venous blood sample collection in order to assess:
  -Malondialdehyde (MDA) is one of the final products of polyunsaturated fatty acids peroxidation in the cells. An increase in free radicals causes overproduction of MDA. Malondialdehyde level is commonly known as a marker of oxidative stress and the antioxidant status in cancerous patients: normal level is.120 nM (SD 36.26)
The NOD-like receptor family protein 3 (ng /ml) | 6 months
  This is by venous blood sample collection in order to assess:
  -The NOD-like receptor family protein 3 (Serum NLRP-3 inflammasome): NR is 2.65 (ng /ml), The NLRP3 inflammasome is considered to be a main pathway for proinflammatory cytokine release in the liver and is strongly involved in the pathogenesis of the liver fibrogenesis
Serum cytokeratin-18 (U/L) | 6 months
  This is by venous blood sample collection in order to assess:
  -Serum cytokeratin-18 the normal range is between 68 to 3000 U/L CK-18 levels increase as the mean of NASH CK18 is present in huge amount in liver. It is an intermediate filament protein representing 5% of the hepatic proteins.

SECONDARY OUTCOMES:
Adverse effects of the intervening drugs | 6 months
  Adverse effects:
  -Any side effects will be reported and graded according to common terminology criteria for adverse events version 5.00 (CTCAE).
  Drug- Drug interactions
  * Any potential drug interactions between administered drugs will be monitored for each patient and corrective actions will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Mohammed Hussein, Assis.Prof, Study Chair — Beni-Suef University; Mona Ahmed Emam, Lecturer, Study Director — Beni-Suef University; Hasnaa Osama Hamed, Lecturer, Study Director — Beni-Suef University
Locations (1):
- Tanta university hospital, Tanta, Gharbyia, Egypt

REFERENCES:
- [Background] El Hadi H, Vettor R, Rossato M. Vitamin E as a Treatment for Nonalcoholic Fatty Liver Disease: Reality or Myth? Antioxidants (Basel). 2018 Jan 16;7(1):12. doi: 10.3390/antiox7010012. PMID 29337849
- [Background] Venetsanaki V, Karabouta Z, Polyzos SA. Farnesoid X nuclear receptor agonists for the treatment of nonalcoholic steatohepatitis. Eur J Pharmacol. 2019 Nov 15;863:172661. doi: 10.1016/j.ejphar.2019.172661. Epub 2019 Sep 16. PMID 31536725
- [Background] Basaranoglu M, Basaranoglu G, Senturk H. From fatty liver to fibrosis: a tale of "second hit". World J Gastroenterol. 2013 Feb 28;19(8):1158-65. doi: 10.3748/wjg.v19.i8.1158. PMID 23483818
- [Background] Tzanaki I, Agouridis AP, Kostapanos MS. Is there a role of lipid-lowering therapies in the management of fatty liver disease? World J Hepatol. 2022 Jan 27;14(1):119-139. doi: 10.4254/wjh.v14.i1.119. PMID 35126843
- [Background] Ioannou GN, Van Rooyen DM, Savard C, Haigh WG, Yeh MM, Teoh NC, Farrell GC. Cholesterol-lowering drugs cause dissolution of cholesterol crystals and disperse Kupffer cell crown-like structures during resolution of NASH. J Lipid Res. 2015 Feb;56(2):277-85. doi: 10.1194/jlr.M053785. Epub 2014 Dec 17. PMID 25520429
- [Background] Ahsan F, Oliveri F, Goud HK, Mehkari Z, Mohammed L, Javed M, Althwanay A, Rutkofsky IH. Pleiotropic Effects of Statins in the Light of Non-Alcoholic Fatty Liver Disease and Non-Alcoholic Steatohepatitis. Cureus. 2020 Sep 14;12(9):e10446. doi: 10.7759/cureus.10446. PMID 33072455
- [Background] Schierwagen R, Maybuchen L, Hittatiya K, Klein S, Uschner FE, Braga TT, Franklin BS, Nickenig G, Strassburg CP, Plat J, Sauerbruch T, Latz E, Lutjohann D, Zimmer S, Trebicka J. Statins improve NASH via inhibition of RhoA and Ras. Am J Physiol Gastrointest Liver Physiol. 2016 Oct 1;311(4):G724-G733. doi: 10.1152/ajpgi.00063.2016. Epub 2016 Sep 15. PMID 27634010
- [Background] Kargiotis K, Katsiki N, Athyros VG, Giouleme O, Patsiaoura K, Katsiki E, Mikhailidis DP, Karagiannis A. Effect of rosuvastatin on non-alcoholic steatohepatitis in patients with metabolic syndrome and hypercholesterolaemia: a preliminary report. Curr Vasc Pharmacol. 2014 May;12(3):505-11. doi: 10.2174/15701611113119990009. PMID 24805248
- [Background] Antonopoulos S, Mikros S, Mylonopoulou M, Kokkoris S, Giannoulis G. Rosuvastatin as a novel treatment of non-alcoholic fatty liver disease in hyperlipidemic patients. Atherosclerosis. 2006 Jan;184(1):233-4. doi: 10.1016/j.atherosclerosis.2005.08.021. Epub 2005 Oct 5. No abstract available. PMID 16168995
- [Background] Gentric G, Maillet V, Paradis V, Couton D, L'Hermitte A, Panasyuk G, Fromenty B, Celton-Morizur S, Desdouets C. Oxidative stress promotes pathologic polyploidization in nonalcoholic fatty liver disease. J Clin Invest. 2015 Mar 2;125(3):981-92. doi: 10.1172/JCI73957. Epub 2015 Jan 26. PMID 25621497
- [Background] Hutcheson R, Rocic P. The metabolic syndrome, oxidative stress, environment, and cardiovascular disease: the great exploration. Exp Diabetes Res. 2012;2012:271028. doi: 10.1155/2012/271028. Epub 2012 Jul 9. PMID 22829804
- [Background] Ore A, Akinloye OA. Oxidative Stress and Antioxidant Biomarkers in Clinical and Experimental Models of Non-Alcoholic Fatty Liver Disease. Medicina (Kaunas). 2019 Jan 24;55(2):26. doi: 10.3390/medicina55020026. PMID 30682878
- [Background] Van Herck MA, Weyler J, Kwanten WJ, Dirinck EL, De Winter BY, Francque SM, Vonghia L. The Differential Roles of T Cells in Non-alcoholic Fatty Liver Disease and Obesity. Front Immunol. 2019 Feb 6;10:82. doi: 10.3389/fimmu.2019.00082. eCollection 2019. PMID 30787925
- [Background] de Andrade KQ, Moura FA, dos Santos JM, de Araujo OR, de Farias Santos JC, Goulart MO. Oxidative Stress and Inflammation in Hepatic Diseases: Therapeutic Possibilities of N-Acetylcysteine. Int J Mol Sci. 2015 Dec 18;16(12):30269-308. doi: 10.3390/ijms161226225. PMID 26694382
- [Background] Dludla PV, Nkambule BB, Mazibuko-Mbeje SE, Nyambuya TM, Marcheggiani F, Cirilli I, Ziqubu K, Shabalala SC, Johnson R, Louw J, Damiani E, Tiano L. N-Acetyl Cysteine Targets Hepatic Lipid Accumulation to Curb Oxidative Stress and Inflammation in NAFLD: A Comprehensive Analysis of the Literature. Antioxidants (Basel). 2020 Dec 16;9(12):1283. doi: 10.3390/antiox9121283. PMID 33339155
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Derived] Zakaria AY, Badawi R, Osama H, Abdelrahman MA, El-Kalaawy AM. New Approach Combination-Dosed Therapy for Nonalcoholic Steatohepatitis Versus Vitamin E: A Randomized Controlled Trial. Clin Ther. 2025 Aug;47(8):e19-e30. doi: 10.1016/j.clinthera.2025.05.006. Epub 2025 Jun 6. PMID 40480879
- [Derived] Zakaria AY, Badawi R, Osama H, Abdelrahman MA, El-Kalaawy AM. A Comparative Study of N-Acetyl Cysteine, Rosuvastatin, and Vitamin E in the Management of Patients with Non-Alcoholic Steatohepatitis: A Randomized Controlled Trial. Pharmaceuticals (Basel). 2025 Apr 29;18(5):650. doi: 10.3390/ph18050650. PMID 40430469